CLINICAL TRIAL: NCT05387707
Title: A Two-part, Multicenter, Randomized, Double-blind Study to Evaluate the Efficacy and Safety of Oral Difelikefalin as Adjunct Therapy to a Topical Corticosteroid for Moderate-to-Severe Pruritus in Adult Subjects With Atopic Dermatitis
Brief Title: Study to Evaluate the Efficacy and Safety of Oral Difelikefalin as Adjunct Therapy to a Topical Corticosteroid for Moderate to Severe Pruritus in Subjects With Atopic Dermatitis
Acronym: KIND-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: In Part A of the study, oral difelikefalin as adjunct to topical corticosteroids (TCS) did not demonstrate meaningful clinical benefit compared to TCS alone.
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR845-310501
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Pruritus; Atopic Dermatitis
Keywords: Atopic Dermatitis; Pruritus; CR845; Chronic Itch; difelikefalin; Itch; Itching; Generalized pruritus; Eczema
MeSH Terms: conditions — Pruritus; Dermatitis, Atopic; Eczema | interventions — difelikefalin

STUDY DESIGN:
Intervention Model Description: Part A includes 4 arms and Part B includes 2 arms.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Difelikefalin 0.25 mg tablets plus TCS cream (Experimental): Oral difelikefalin tablets administered twice daily. TCS cream applied by study subjects to skin lesions once a day until control is achieved, then as needed.
  Interventions: Drug: difelikefalin 0.25 mg; Drug: TCS Cream
- Difelikefalin 0.5 mg tablets plus TCS cream (Experimental): Oral difelikefalin tablets administered twice daily. TCS cream applied by study subjects to skin lesions once a day until control is achieved, then as needed.
  Interventions: Drug: difelikefalin 0.5 mg; Drug: TCS Cream
- Placebo tablets plus TCS cream (Active Comparator): Oral placebo tablets administered twice daily. TCS cream applied by study subjects to skin lesions once a day until control is achieved, then as needed
  Interventions: Drug: TCS Cream; Drug: Placebo
- Placebo tablets plus Vehicle cream (Part A only) (Placebo Comparator): Oral placebo tablets administered twice daily. Vehicle cream applied by study subjects to skin lesions once a day until control is achieved, then as needed
  Interventions: Drug: Placebo; Drug: Vehicle Cream

INTERVENTIONS:
Drug: difelikefalin 0.25 mg — Oral difelikefalin 0.25 mg tablets administered twice daily
  Other Names: CR845
  Arms: Difelikefalin 0.25 mg tablets plus TCS cream
Drug: difelikefalin 0.5 mg — Oral difelikefalin 0.5 mg tablets administered twice daily
  Other Names: CR845
  Arms: Difelikefalin 0.5 mg tablets plus TCS cream
Drug: TCS Cream — TCS cream applied by study subjects to skin lesions once a day until control is achieved, then as needed
  Arms: Difelikefalin 0.25 mg tablets plus TCS cream; Difelikefalin 0.5 mg tablets plus TCS cream; Placebo tablets plus TCS cream
Drug: Placebo — Oral Placebo tablets administered twice daily
  Arms: Placebo tablets plus TCS cream; Placebo tablets plus Vehicle cream (Part A only)
Drug: Vehicle Cream — Vehicle Cream applied by study subjects to skin lesions once a day until control is achieved, then as needed
  Arms: Placebo tablets plus Vehicle cream (Part A only)

SUMMARY:
This is a two-part, multicenter, randomized, double-blind study to evaluate the efficacy and safety of oral difelikefalin as adjunct therapy to a topical corticosteroid (TCS) for moderate-to-severe pruritus in adult subjects with atopic dermatitis (AD).

DETAILED DESCRIPTION:
Part A of this study includes a 12-week Double-blind Treatment Period and a 52-week Open-label Extension Period. Subjects will be randomized to receive oral difelikefalin 0.25 mg tablets BID plus TCS cream, difelikefalin 0.5 mg tablets BID plus TCS cream, placebo tablets BID plus TCS cream or placebo tablets BID plus vehicle cream.

Part B of this study includes a 12-week Double-blind Treatment Period and 52-week Open-label Extension Period. Subjects will be randomized to receive oral difelikefalin 0.25 mg or 0.5 mg tablets BID plus TCS cream or oral placebo tablets BID plus TCS cream. Part A results at week 12 will inform Part B.

Subjects who participated in Part A of the study may not participate in Part B.

All subjects will sign an informed consent form (ICF) and undergo screening for study eligibility.

ELIGIBILITY:
Key Inclusion Criteria:

To be eligible for inclusion into the study, a patient must meet the following criteria:

* Subject has clinically confirmed diagnosis of active AD;
* Subject has chronic pruritus related to AD;
* Subject has moderate to severe pruritus;
* Female subject is not pregnant or nursing during any period of the study.

Key Exclusion Criteria:

A patient will be excluded from the study if any of the following criteria are met:

* Subject has clinically infected AD;
* Subject has pruritus attributed to a cause other than AD;
* Subject has any clinically significant medical condition or physical/laboratory/ECG/vital signs abnormality that would, in the opinion of the investigator, put the subject at undue risk or interfere with interpretation of study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving an improvement from baseline ≥4 points with respect to the weekly mean of the daily 24-hour I-NRS score at Week 12 | Week 12

SECONDARY OUTCOMES:
Proportion of subjects achieving ≥ 4 point improvement from baseline in the weekly mean of the daily 24-hour I-NRS score at Week 4 | Week 4
Proportion of subjects with ≥ 3 point improvement from baseline in the weekly mean of the daily 24-hour Sleep Disturbance NRS score at the end of Week 12 (among subjects with a Sleep Disturbance NRS score of > 3 at baseline) | Week 12
Proportion of subjects achieving ≥ 4 point improvement from baseline in the weekly mean of the daily 24-hour I-NRS score at Week 2 | Week 2
Proportion of subjects achieving ≥ 4 point improvement from baseline in the weekly mean of the daily 24-hour I-NRS score at Week 1 | Week 1
Mean change and mean percent change from baseline in EASI score at Week 12. | Week 12
Proportion of subjects achieving a vIGA-ADTM score of clear (0) or almost clear (1) with a 2-point improvement from baseline at Week 12 (among subjects with a vIGA-ADTM score ≥ 3 at Day 1) | Week 12
Proportion of subjects achieving a vIGA-ADTM score of clear (0) or almost clear (1) with a 2-point improvement from baseline at Week 12 (among subjects with a vIGA-ADTM score ≥ 2 at Day 1) | Week 12
Proportion of subjects achieving at least ≥ 3-point improvement in the Skin Pain NRS score at Week 12 (among subjects with a Skin Pain NRS score > 3 at Day 1) | Week 12
Proportion of subjects with ≥ 4 point improvement from baseline in Dermatology Life Quality Index (DLQI) score at Week 12 (among subjects with DLQI score > 4 at baseline) | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Cara Therapeutics, Study Director — Cara Therapeutics
Locations (60):
- United States (60):
  - Cara Therapeutics Study Site, Scottsdale, Arizona
  - Cara Therapeutics Study Site, Fort Smith, Arkansas
  - Cara Therapeutics Study Site, Rogers, Arkansas
  - Cara Therapeutics Study Site, Fountain Valley, California
  - Cara Therapeutics Study Site, Lomita, California
  - Cara Therapeutics Study Site, Los Angeles, California
  - Cara Therapeutics Study Site, Redwood City, California
  - Cara Therapeutics Study Site, Sacramento, California
  - Cara Therapeutics Study Site, San Diego, California
  - Cara Therapeutics Study Site 2, Santa Monica, California
  - Cara Therapeutics Study Site, Santa Monica, California
  - Cara Therapeutics Study Site, Valencia, California
  - Cara Therapeutics Study Site, Denver, Colorado
  - Cara Therapeutics Study Site, Brandon, Florida
  - Cara Therapeutics Study Site, Coral Gables, Florida
  - Cara Therapeutics Study Site, Delray Beach, Florida
  - Cara Therapeutics Study Site, Hollywood, Florida
  - Cara Therapeutics Study Site, North Miami Beach, Florida
  - Cara Therapeutics Study Site, Orlando, Florida
  - Cara Therapeutics Study Site, Saint Augustine, Florida
  - Cara Therapeutics Study Site, St. Petersburg, Florida
  - Cara Therapeutics Study Site, Sweetwater, Florida
  - Cara Therapeutics Study Site, Tampa, Florida
  - Cara Therapeutics Study Site, Marietta, Georgia
  - Cara Therapeutics Study Site, Indianapolis, Indiana
  - Cara Therapeutics Study Site, Plainfield, Indiana
  - Cara Therapeutics Study Site, South Bend, Indiana
  - Cara Therapeutics Study Site, Overland Park, Kansas
  - Cara Therapeutics Study Site, Louisville, Kentucky
  - Cara Therapeutics Study Site, Baton Rouge, Louisiana
  - Cara Therapeutics Study Site, Houma, Louisiana
  - Cara Therapeutics Study Site, Metairie, Louisiana
  - Cara Therapeutics Study Site, New Orleans, Louisiana
  - Cara Therapeutics Study Site, Rockville, Maryland
  - Cara Therapeutics Study Site, Brighton, Massachusetts
  - Cara Therapeutics Study Site, Auburn Hills, Michigan
  - Cara Therapeutics Study Site, Clinton Township, Michigan
  - Cara Therapeutics Study Site, Detroit, Michigan
  - Cara Therapeutics Study Site, Waterford, Michigan
  - Cara Therapeutics Study Site, Hackensack, New Jersey
  - Cara Therapeutics Study Site, Huntersville, North Carolina
  - Cara Therapeutics Study Site, Raleigh, North Carolina
  - Cara Therapeutics Study Site, Athens, Ohio
  - Cara Therapeutics Study Site, Bexley, Ohio
  - Cara Therapeutics Study Site, Boardman, Ohio
  - Cara Therapeutics Study Site, Oklahoma City, Oklahoma
  - Cara Therapeutics Study Site, Philadelphia, Pennsylvania
  - Cara Therapeutics Study Site, Plymouth Meeting, Pennsylvania
  - Cara Therapeutics Study Site, Sugarloaf, Pennsylvania
  - Cara Therapeutics Study Site, Charleston, South Carolina
  - Cara Therapeutics Study Site, Knoxville, Tennessee
  - Cara Therapeutics Study Site, Thompson's Station, Tennessee
  - Cara Therapeutics Study Site, Arlington, Texas
  - Cara Therapeutics Study Site, Austin, Texas
  - Cara Therapeutics Study Site, Bellaire, Texas
  - Cara Therapeutics Study Site, Houston, Texas
  - Cara Therapeutics Study Site, San Antonio, Texas
  - Cara Therapeutics Study Site, Springville, Utah
  - Cara Therapeutics Study Site, Spokane, Washington
  - Cara Therapeutics Study Site, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No